CLINICAL TRIAL: NCT00652652
Title: Evaluation of Synergy Between Natrecor and Furosemide on Renal and Neurohormone Responses in Chronic Heart Failure: A Phase-IV Study
Brief Title: Evaluation of Combined Action Between Natrecor and Furosemide on Kidney and Neurohormone Responses in Chronic Heart Failure: A Phase-IV study704.351 / DSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR003319
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Congestive Heart Failure; Chronic Heart Failure
Keywords: Congestive Heart Failure (CHF); Heart Failure; Chronic Heart Failure; Dyspnea; nesiritide; Natrecor
MeSH Terms: conditions — Heart Failure; Dyspnea | interventions — Natriuretic Peptide, Brain; Furosemide

INTERVENTIONS:
Drug: nesiritide, furosemide

SUMMARY:
This is a randomized, open-label, three-way crossover design study with 3 treatment groups:TREATMENT A: Furosemide;TREATMENT B: Nesiritide administered IV bolus, followed by an infusion for 6 hours;TREATMENT C: Treatment B for at least 15 minutes, then administration of treatment AAll sequences involving both furosemide and nesiritide had the nesiritide infusion started first, at least 15 minutes before furosemide was administered. Each treatment will be administered according to 1 of 6 sequences to which patients are randomized. Patients will remain in the Clinical Research Unit for 7 days, with treatments administered on Days 2, 4, and 6, with equilibrium (rest) days on Days 1, 3, and 5. All patients will be followed for safety throughout the treatment phase, and by telephone between 7 and 14 days after they are discharged from the Clinical Research Unit.

DETAILED DESCRIPTION:
Nesiritide is the recombinant form of human B-type natriuretic peptide (hBNP). The drug is indicated for the IV treatment of patients with acutely decompensated congestive heart failure who have shortness of breath at rest or with minimal activity. hBNP has been found to have favorable effects on the hemodynamic profile of patientswith heart failure, producing a dose-dependent fall in systemic vascular resistance (SVR) and a mild reduction in arterial pressure. Furosemide (Lasix) is frequently administered to patients with acutely decompensated heart failure to relieve pulmonary vascular congestion and promote diuresis. The efficacy of furosemide is based on its ability to markedly enhance sodium excretion and decrease intravascular volume despite the presence of decreased renal perfusion pressure. However, furosemide is associated with a variety of deleterious effects and, by itself, may not consistently cause diuresis or natriuresis. The administration of intravenous (IV) furosemide causes a slight increase in mean arterial pressure and systemic vascular resistance and a decrease in cardiac output before the onset of diuresis in patients with heart failure. This results in alterations in renal blood flow and a decrease in glomerular filtration rate (GFR). These effects are related to the activation of the renin angiotensin-aldosterone (RAA) systemIn addition, the plasma norepinephrine level increases acutely after administration of IV furosemide. Chronic use of furosemide further aggravates the sympathetic nervous system (SNS) and RAA activation due to relative reductions in intravascular volume. In previous studies of patients with congestive heart failure (CHF), nesiritide increased natriuresis and diuresis while maintaining or increasing GFR. Additionally, hBNP has produced neuroendocrinologic alterations including decreased aldosterone levels and a mild decrease in peripheral renin activity. Therefore, nesiritide may inhibit the anti-natriuretic effect of angiotensin II and aldosterone on proximal and distal tubules of the kidney. Given the contrasting properties of furosemide and nesiritide on neuroendocrine activation in the setting of heart failure, the combination of these agents may be synergistic. Nesiritide may reduce the mild acute vasoconstrictor and neuroendocrinologic properties of furosemide while augmenting its diuretic and natriuretic effects. This trial is a randomized, open-label, three-way crossover design study. The patient population will consist of patients with symptomatic CHF (New York Heart Association [NYHA] Class II or III). All patients are to receive all 3 of the following treatments, administered in randomized order. TREATMENT A: Furosemide administered as a 40 mg IV bolus over 2 minutes. TREATMENT B: Nesiritide administered as a 2 mcg/kg IV bolus, followed by an infusion of 0.01 mcg/kg/min for 6 hours. TREATMENT C: Treatment B for at least 15 minutes, then administration of treatment A. Each of the treatments will be administered according to 1 of the 6 sequences to which patients are randomized. Each treatment will be followed by a 1-day equilibrium period. Efficacy will be assessed by the evaluation of urinary excretion rate of sodium, urinary flow rate, urinary excretion of potassium, calcium and magnesium, urinary excretion of cGMP and furosemide, change from baseline in plasma aldosterone, change in BNP levels and iohexol clearance (Glomerular Filtration Rate). Safety will be assessed through out the study by way of physical examinations and evaluation of daily blood chemistries, adverse events (AEs), and serious adverse events (SAEs). TREATMENT A: Furosemide administered as a 40 mg intravenous (IV) bolus over 2 minutesTREATMENT B: Nesiritide administered as a 2 mcg/kg IV bolus, followed by an infusion of 0.01 mcg/kg/min for 6 hoursTREATMENT C: Treatment B for at least 15 minutes, then administration of treatment A

ELIGIBILITY:
Inclusion Criteria:

* Chronic symptomatic NYHA Class II or III CHF for at least 90 days before the study
* Left ventricular systolic dysfunction as evidenced by left ventricular ejection fraction < 40%, measured using contrast or radionuclide ventriculography or by echocardiography, within 180 days of the study start
* Serum potassium > 3.5 mEq/L.
* Chronic oral daily requirement of 80-240 mg of furosemide for at least 7 days before the study start
* Receiving a stable medical regimen for CHF for at least 60 days before the study start, including angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARBs), and/or beta-blockers.

Exclusion Criteria:

* Clinical instability such that withholding diuretic therapy would be unsafe
* Significant renal impairment (e.g., creatinine clearance < 45 mL/min by the Cockcroft-Gault formula), or changing renal function during the 7 days before study start, or intrinsic renal disease
* Systolic blood pressure (SBP) consistently < 90 mm Hg
* Myocardial infarction within 90 days of study start, unstable angina within 14 days of study start, or any clinical evidence of active myocardial ischemia
* Percutaneous coronary intervention or cardiac surgery within 90 days of study start
* Restrictive or obstructive cardiomyopathy, constrictive pericarditis, pericardial tamponade, other conditions in which cardiac output was dependent on venous return, or for subjects expected to have low filling pressures
* Prior cardiac or renal allografts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Patient's urinary excretion rate of sodium

SECONDARY OUTCOMES:
Patient's urinary flow rate, urinary excretion of potassium, calcium and magnesium, and urinary excretion of cGMP and furosemide

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- See also: Evaluation of combined action Between Natrecor and Furosemide on Kidney and Neurohormone Responses in Chronic Heart failure: A Phase-IV study704.351 / DSS — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=953&filename=CR003319_CSR.pdf